CLINICAL TRIAL: NCT02404519
Title: Intervention Study on the Effect of Vitamin K2 (Menaquinone-7) Supplementation on the Vascular Stiffness in Subjects With Poor Vitamin K-status
Brief Title: Vitamin K2 Effect on Vascular Stiffening in Subjects With a Poor Vitamin K-status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Marjo Knapen, Marjo Knapen, BSc, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC143058
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Vascular Stiffness
Keywords: Vitamin K; Menaquinone-7; Matrix Gla Protein; Vascular stiffness
MeSH Terms: interventions — menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menaquinone-7 (Active Comparator): Menaquinone-7 180 microgram tablet, by mouth, daily for 1 year
  Interventions: Dietary Supplement: Menaquinone-7
- Placebo (Placebo Comparator): Placebo tablet, by mouth, daily for 1 year
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Menaquinone-7 — 1 tablet containing 180 micrograms MK-7 taken orally every day during 1 year
  Other Names: MK-7
  Arms: Menaquinone-7
Dietary Supplement: Placebo — 1 tablet without MK-7 taken orally every day during 1 year
  Arms: Placebo

SUMMARY:
Vitamin K is required for the activation of the inhibitor of vascular calcification: Matrix Gla Protein (MGP). In an earlier study the beneficial effect of menaquinone-7 (MK-7), a vitamin K2 form, was observed on the stiffness of the vessel wall in postmenopausal women. It decreased the circulating form of inactive MGP and improved the vascular elasticity (local) and aortic pulse wave velocity (regional). The decrease of circulating inactive MGP was observed after 2-3 months MK-7 supplementation and the effect of MK-7 on the clinical endpoints was observed within 3 years of supplementation. It is demonstrated in several studies that cardiovascular risk increases with decreasing vitamin K intake and increasing levels of inactive MGP. In this study the investigators select subjects in the highest tertile of circulating inactive MGP. This study group will consist of subjects with increased cardiovascular risk and it is expected that effects of MK-7 on clinical endpoints in this group will be measurable within 1 year of supplementation.

Vascular stiffness can be determined with different techniques. The vascular characteristics determined with Pulse Wave Velocity (PWV), ultrasound of the common carotid artery and accelerated plethysmography (APG) with a fingertip device will be compared in a follow-up study.

DETAILED DESCRIPTION:
This study will be a double-blind randomized placebo-controlled intervention study. In total 240 healthy men and women between 40 and 70 years will be recruited in the province of Limburg through small advertisements in local newspapers.

Eligible participants will be randomized into 2 study groups:

* Group 1: MK-7 (1 tablet: MK-7 dosage is 180 μg)
* Group 2: Placebo (1 tablet: MK-7 dosage is 0 µg) Each group will consist of 120 participants. A double-blind design is chosen to avoid the occurrence of bias during the study. After randomization, the participants consume the placebo or MK-7 tablets once daily with either breakfast or dinner during one year.

People who are interested to participate will come to the research laboratory of VitaK for a screening visit (day -14). During this visit, the investigator will check whether the volunteers are eligible for inclusion based on the in- and exclusion criteria. After meeting the inclusion criteria and none of the exclusion criteria, volunteers will be assigned a randomization number from a computer-generated randomization list. A stratified block randomization will be performed for gender, in order to avoid unequal distribution of men and women among the 2 treatment groups.

On-site measurements will be performed at t=0 and after 1 year of treatment: the carotid-femoral Pulse Wave Velocity (cfPWV; primary outcome) and echotracking of the common carotid artery to assess the vascular stiffness (secondary outcome). A Whole Body scan with DXA will be performed to determine total fat and lean mass of the participants. Blood will be taken after an overnight fasting period at t=0 and after 1 year to measure the circulating level of inactive MGP.

Results from our previous study (NCT00642551) showed significant changes in vascular characteristics, pulse wave velocity after a 3 year intervention period with a daily dosage of 180 µg MK-7 in 240 postmenopausal women. After 1 year MK-7 intervention inactive MGP levels (improvement of vascular vitamin K status) were decreased 50% compared to placebo and remained at this level during the following 2 years of intervention.

Recently published population-based studies show that the unfavorable cardiovascular outcomes are mainly attributable to those within the highest quartile of circulating dp-ucMGP. We expect, therefore, that an intervention study among preselected subjects with poor vascular vitamin K status (inactive MGP levels > 400 pmol/L) and treatment with the same dosage MK-7 (i.e. 180 µg/day) during one year will have a more pronounced effect on arterial stiffening and pulse wave velocity.

The follow-up study will be performed at the end of the intervention period of 1 year, with participants who have completed the one year intervention study. From this study population eligible participants (men and women) will be selected. In total 100 participants will be invited. Measurements will be performed at the same day: the carotid-femoral Pulse Wave Velocity (cfPWV), echotracking of the common carotid artery to assess the vascular stiffness and accelerated plethysmography measurements (APG) will be assessed using an fingertip oximeter StiffnoGraph (Taiwan): heart rate, SpO2 (oxygen saturation) and stiffness score.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 40 and 70 years old
* Subjects with body weight and height according to BMI between 20 and 35 kg/m2
* Subjects of Caucasian race
* Subject has given written consent to take part in the study
* Subjects with circulating dp-ucMGP higher than 400 pmol/L

Exclusion Criteria:

* Subjects with cardiovascular disease
* Subjects with hyperlipidaemia
* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Use of more than 3 units alcohol/day
* Subjects receiving oestrogen treatment (women)
* Subjects using corticosteroids
* Subjects using oral anticoagulants and subjects with clotting disorders
* Subjects using vitamin K containing multivitamins or supplements

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline carotid-femoral Pulse Wave Velocity (PWV) at 1 year | 1 year
  PWV (in m/s) will be assessed noninvasively by measuring carotid-femoral PWV, using mechanotransducers applied directly on the skin.

SECONDARY OUTCOMES:
Change from baseline diameter of the common carotid artery at 1 year | 1 year
  The diameter of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The diameter will be assessed in mm.
Diameter of the common carotid artery | up to 1 year post-intervention
  The diameter of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The diameter will be assessed in mm.
Change from baseline distension of the common carotid artery at 1 year | 1 year
  The distension of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The distension will be assessed in micrometer.
Distension of the common carotid artery | up to 1 year post-intervention
  The distension of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The distension will be assessed in micrometer.
Change from baseline intima-media thickness (IMT) of the common carotid artery at 1 year | 1 year
  The IMT of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The IMT will be assessed in micrometer.
Intima-media thickness (IMT) of the common carotid artery | up to 1 year post-intervention
  The IMT of the common carotid artery will be measured using a linear array transducer connected to an ultrasound scanner. The IMT will be assessed in micrometer.
circulating inactive Matrix Gla Protein (dp-ucMGP) | baseline and 1 year
  Dp-ucMGP (in pM) will be measured using a sandwich ELISA, based on monoclonal antibodies.
carotid-femoral Pulse Wave Velocity (PWV) | up to 1 year post-intervention
  PWV (in m/s) will be assessed noninvasively by measuring carotid-femoral PWV, using mechanotransducers applied directly on the skin.

OTHER OUTCOMES:
Follow-up study outcome: Accelerated phlethysmography (APG) | Up to 1 year post-intervention
  Accelerated plethysmography measurements will be assessed using an fingertip oximeter indicating Stiffness Score 1 through 6.

CONTACTS AND LOCATIONS:
Overall Officials: Marjo HJ Knapen, BSc, Principal Investigator — VitaK BV/Maastricht University